CLINICAL TRIAL: NCT06388707
Title: A Prospective, Open-label, Single-arm, Multi-center, Pilot Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Low-intensity Focused Ultrasound Neuromodulation in Patients With Drug-resistant Unilateral or Bilateral Temporal Lobe Epilepsy
Brief Title: A Safety, Tolerability, and Preliminary Efficacy of Low-intensity Focused Ultrasound Neuromodulation in Patients With Drug-resistant Epilepsy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NaviFUS Corporation (Industry)
Collaborators: NaviFUS US LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NF-2022-01
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Drug Resistant Epilepsy; Epilepsy
Keywords: NaviFUS System; Focused Ultrasound; Low-Intensity Focused Ultrasound
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FUS treatment (Experimental)
  Interventions: Device: NaviFUS System

INTERVENTIONS:
Device: NaviFUS System — FUS treatment will be conducted with following exposure parameters: intracranial spatial-peak temporal-average intensity (ISPTA) ceiling level: 2.8 W/cm2, burst length: 3 ms, duration: max. three consecutive 10-minute FUS exposures with two 5-minute intermission intervals.

SUMMARY:
This will be a prospective, open-label, single-arm, multi-center, pilot study to evaluate the safety, tolerability, and preliminary efficacy of low-intensity focused ultrasound (LIFU) neuromodulation using NaviFUS System in patients with drug-resistant unilateral or bilateral temporal lobe epilepsy (DR-TLE).

DETAILED DESCRIPTION:
The study aims to demonstrate the safety and preliminary efficacy of LIFU neuromodulation in DR-TLE patients, showing its ability to decrease targeted neuronal activity and alleviate epileptic seizures.

Patients diagnosed with epilepsy who meet all eligibility criteria may participate in this study by providing informed consent, either in person or through their legal representative. Eligible patients will undergo a 2-month baseline observation screening period and will be asked to keep a 8-week seizure diary. This diary will serve as a baseline prior to treatment and will continue to be recorded throughout the treatment and follow-up period.

This study will enroll a maximum of 8 eligible patients through competitive enrollment. Patients will receive a total of 6 FUS treatments over 3 consecutive weeks using assigned ultrasound exposure doses generated by the NaviFUS System. Following treatment, there will be a 12-week follow-up period. Patients will be allowed concomitant use of anti-seizure medications (ASMs) throughout the whole study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age at the time of enrollment.
2. Patients with drug-resistant temporal lobe epilepsy (DR-TLE), defined as failure of adequate trials of two tolerated, appropriately chosen and used anti-epileptic drug schedules (whether as monotherapies or in combination).
3. Focal-onset seizures with or without secondary generalization and no more than two known seizure onset zones (seizure foci), at least one which is in the mesial temporal lobe.
4. At least 4 focal-onset seizures with objectively visible or significantly disabling manifestations in the 8-week baseline and at least one seizure per month in the baseline.
5. MRI and EEG within the past 3 years. At least one prior EEG should demonstrate interictal or ictal focal epileptiform findings.
6. Patients with the central of FUS exposure region are located at least 30 mm distance beneath the skull bone.
7. Patients must be on a stable regimen of anti-epileptic drugs (AEDs) for at least 30 days at the time of enrollment, except for rescue benzodiazepines or occasional extra doses of ongoing medicines, as required.
8. Females of childbearing potential must have a negative pregnancy test prior to the first treatment. Females of childbearing potential and male patients with a partner of childbearing potential must agree to follow acceptable method of contraception (as outlined below) from prior to the first study treatment to 3 months after the last study treatment. Standard acceptable methods include use of highly effective method of contraception, including: hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom, spermicide, vasectomy, intrauterine device, and abstinence from sex.
9. Patients are able and willing to have their hair shaved in the region where the coupling membrane will touch (or if they prefer, whole head).
10. Patients are able to complete all clinical trial-related questionnaires in English, including with the use of a suitable interpreter.
11. Patients or their legal representatives are able to provide written informed consent for participation in the trial and comply with study requirements in the opinion of the Investigator during the study period.

Exclusion Criteria:

1. Patients who have primary generalized epilepsy, mixed focal and generalized epilepsy, or any history of non-epileptic seizures.
2. Patients who have experienced tonic-clonic status epilepticus in the 12 months before the time of enrollment in the study. Subjects with focal status epilepticus may be considered at the discretion of the Investigator.
3. The only feasible sonication pathway to the seizure onset zones involves either:

   1. Skull area is covered by previous surgical site(s), scars, scalp disorders (e.g., eczema, psoriasis), or scalp atrophy.
   2. Clips or other metallic implanted objects in the skull or brain, except shunts.
   3. A prior craniotomy site.
4. Patients with a potentially acute or progressive neurologic disorder (e.g., brain tumor, multiple sclerosis, dementia, or intracranial vascular lesion).
5. Implanted electronic device, for example, implanted cardioverter-defibrillator (ICD), cardiac pacemaker, permanent medication pumps, cochlear implants, responsive neurostimulator, deep brain stimulation (DBS), or other electronic devices implanted in the brain. If a patient has a working Vagus Nerve Stimulator (VNS) in place, the settings should remain stable throughout the trial and the device will be turned off prior to each sonication treatment and then turned back on afterward.
6. Patients with severe depression, active suicidal ideation or behavior (as per the C-SSRS), active psychosis (excluding time-limited postictal psychosis), or psychiatric hospitalization in the year before time of enrollment.
7. Patient has an IQ < 70, based on the Wechsler Abbreviated Scale of Intelligence (WASI-II or other Wechsler IQ measure).
8. Coexisting medical problems of sufficient severity to limit compliance with or interpretation of the study.
9. Patients have received an investigational drug or an investigational device within 4 weeks prior to the first treatment.
10. Radiofrequency thermocoagulation (RFTC) within 2 months before time of enrollment.
11. Known history of substance or alcohol abuse within the past year, not counting marijuana.
12. Pregnant or breast-feeding women.
13. Any other condition that, in the Investigator's judgment, might affect study endpoints or might increase the risk to the patients or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | up to 23 weeks
  The incidence and severity of AEs associated with LIFU neuromodulation in patients with drug-resistant unilateral or bilateral temporal lobe epilepsy.

SECONDARY OUTCOMES:
Change from baseline in seizure frequency | up to 23 weeks
  The changes in patient's seizure frequency during and after treatment will be assessed based on the seizure diaries.
Change from baseline in electroencephalography (EEG) epileptiform discharges | up to 15 weeks
  The change in patient's epileptiform discharges after treatment will be assessed based on the EEG recording.
Days of seizure-free | up to 23 weeks
  The changes in number of seizure-free days after FUS treatment(s).
Changes from baseline in Beck Anxiety Inventory (BAI) | up to 23 weeks
  BAI is a 21-question multiple-choice self-report inventory that is used to measure the severity of anxiety. Each answer is scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
Changes from baseline in Beck Depression Inventory (BDI-II) | up to 23 weeks
  BDI-II, a 21-question multiple-choice self-report inventory, is a psychological test used to measure the severity of depression. Each answer is rated on a scale of 0 (none at all) to 3 (severe). Higher total scores indicate more severe depressive symptoms.
Changes from baseline in Personal Impact of Epilepsy Scale (PIES) | up to 23 weeks
  PIES is a 25-item multiple-choice self-report inventory that is used to evaluate the overall impact of seizures, side effects, comorbidities, and overall quality of life for people with epilepsy. Each answer is rated by patient on a scale value of 0 (best) to 4 (worst). Lower total PIES scores reﬂect better overall status.

OTHER OUTCOMES:
Change from baseline in subjective seizure strength | up to 23 weeks
  The changes in patient's seizure strength during and after treatment will be assessed based on the seizure diaries.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Palo Alto, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Virginia School of Medicine, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SG, Tsai CH, Lin CJ, Lee CC, Yu HY, Hsieh TH, Liu HL. Transcranial focused ultrasound pulsation suppresses pentylenetetrazol induced epilepsy in vivo. Brain Stimul. 2020 Jan-Feb;13(1):35-46. doi: 10.1016/j.brs.2019.09.011. Epub 2019 Sep 24. PMID 31575487
- [Background] Chu PC, Yu HY, Lee CC, Fisher R, Liu HL. Pulsed-Focused Ultrasound Provides Long-Term Suppression of Epileptiform Bursts in the Kainic Acid-Induced Epilepsy Rat Model. Neurotherapeutics. 2022 Jul;19(4):1368-1380. doi: 10.1007/s13311-022-01250-7. Epub 2022 May 17. PMID 35581489
- [Background] Lee CC, Chou CC, Hsiao FJ, Chen YH, Lin CF, Chen CJ, Peng SJ, Liu HL, Yu HY. Pilot study of focused ultrasound for drug-resistant epilepsy. Epilepsia. 2022 Jan;63(1):162-175. doi: 10.1111/epi.17105. Epub 2021 Nov 2. PMID 34729772